CLINICAL TRIAL: NCT06461585
Title: Effects of Sprint Interval Training Versus Arabic Exercises BMI Waist-to-hip Ratio and Quality of Life in Obese Women PCOS
Brief Title: Effects of Sprint Interval Training Versus Arabic Exercises BMI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RECRCR&AHS-23-0573
Record Dates: First submitted 2024-06-11; First posted 2024-06-17 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: PCOS
Keywords: BMI; High intensity interval training; PCOS Syndrome; Quality of life
MeSH Terms: interventions — High-Intensity Interval Training; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sprint interval training exercise (Experimental): Group A the Interventional group will receive SIT . Group A will perform SIT 3 times a week for 30-second sprints on a cycle ergometer with 4 minutes of rest between each sprint, complete session will be for 30 -40 minutes.
  Interventions: Other: Sprint interval training
- Arabic exercises (Experimental): Group B will receive the aerobic exercise. Group B will perform the aerobic exercise for 30-40 minutes of moderate-intensity continuous exercise on a treadmill and stationary cycle
  Interventions: Other: Sprint interval training

INTERVENTIONS:
Other: Sprint interval training — Group A the Interventional group will receive SIT . Group A will perform SIT 3 times a week for 30-second sprints on a cycle ergometer with 4 minutes of rest between each sprint, complete session will be for 30 -40 minutes. Group B will receive the aerobic exercise. Group B will perform the aerobic exercise for 30-40 minutes of moderate-intensity continuous exercise on a treadmill and stationary cycle
  Other Names: aerobic exercises

SUMMARY:
Polycystic ovary syndrome (PCOS) is the most common endocrine disorder in women of reproductive age and is the leading cause of infertility and anovulation. According to the Rotterdam criteria, the prevalence of PCOS is estimated to affect up to 20% of the female population. PCOS is characterized by increased androgen production and decreased ovulation leading to clinical manifestations including acne, hirsutism, male pattern baldness, irregular menstrual cycles, and infertility. In addition to concerns about fertility and hyperandrogenism, PCOS is considered a metabolic disorder, with an increased risk of developing insulin resistance (IR), hyperinsulinemia, dyslipidemia, and low-grade inflammation. In addition to genetic involvement, environmental aspects such as obesity conditions. affect the progression of PCOS or even make patients' clinical conditions worse. Exercise is an important component of PCOS management, and exercises have been shown to improve metabolic and reproductive outcomes in women with PCOS. The study will be a randomized clinical trial. This study will be completed in a time duration of 7 months after the approval of the synopsis. Sample size 32 is calculated by the Epi tool.variable for the sample size is BMI. By the non-probability convenience sampling technique, participants will be divided into 2 groups. Group A the Interventional group will receive SIT and Group B will receive the aerobic exercise. Group A will perform SIT 3 times a week for 30-second sprints on a cycle ergometer with 4 minutes of rest between each sprint, complete session will be for 30 -40 minutes while Group B will perform the aerobic exercise for 30-40 minutes of moderate-intensity continuous exercise on a treadmill and stationary cycle. The outcome measure will be evaluated by using the BMI Calculator, PCOSQOL, measuring tape Borg scale. After Collecting data from the before and after treatment sessions. The data will be analyzed by using SPSS version 25.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is the most common endocrine disorder in women of reproductive age and is the leading cause of infertility and anovulation. According to the Rotterdam criteria, the prevalence of PCOS is estimated to affect up to 20% of the female population. PCOS is characterized by increased androgen production and decreased ovulation leading to clinical manifestations including acne, hirsutism, male pattern baldness, irregular menstrual cycles, and infertility. In addition to concerns about fertility and hyperandrogenism, PCOS is considered a metabolic disorder, with an increased risk of developing insulin resistance (IR), hyperinsulinemia, dyslipidemia, and low-grade inflammation. In addition to genetic involvement, environmental aspects such as obesity conditions. affect the progression of PCOS or even make patients' clinical conditions worse. Exercise is an important component of PCOS management, and exercises have been shown to improve metabolic and reproductive outcomes in women with PCOS. The study will be a randomized clinical trial. The study will be conducted in the settings of Jinnah Hospital Lahore, Shapes Gym, and UFC Gym. This study will be completed in a time duration of 7 months after the approval of the synopsis. Sample size 32 is calculated by the Epi tool.variable for the sample size is BMI. By the non-probability convenience sampling technique, participants will be divided into 2 groups. Group A the Interventional group will receive SIT and Group B will receive the aerobic exercise. Group A will perform SIT 3 times a week for 30-second sprints on a cycle ergometer with 4 minutes of rest between each sprint, complete session will be for 30 -40 minutes while Group B will perform the aerobic exercise for 30-40 minutes of moderate-intensity continuous exercise on a treadmill and stationary cycle. The outcome measure will be evaluated by using the BMI Calculator, PCOSQOL, measuring tape Borg scale. After Collecting data from the before and after treatment sessions. The data will be analyzed by using SPSS version 25.

Keywords: Body Mass Index, High-Intensity Interval Training, Polycystic Ovary Syndrome, Quality of Life

ELIGIBILITY:
Inclusion Criteria:

Diagnosed PCOS

* Age: 18 - 35 years.
* BMI ≥25 kg/m2
* Unmarried females (5)
* Oligomenorrhea
* Irregular cycles (Have less than 9 periods in 1 year

Exclusion Criteria:

* Congenital adrenal hyperplasia, androgen-secreting tumors, and Cushing's syndrome
* Cardiovascular diseases and thrombotic diseases.
* Systemic illness (Acute or chronic hepatitis or nephritis, musculoskeletal and pulmonary disorder)
* Taking medications known to affect ovarian function within the past 3 months.
* Patients suffer from mental problems.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female (PCOS)
Enrollment: 36 (Estimated)
Dates: Start 2023-12-10 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-07-10 (Estimated)

PRIMARY OUTCOMES:
Modified Borg CR10 RPE scale (For Exertion level) | 8 weeks
  PCOSQOL
Waist-to-hip ratio: (Measuring tape) | 8 weeks
  BMI Calculator:
  BMI Calculator:

CONTACTS AND LOCATIONS:
Overall Officials: Sabiha Arshad, M.phill, Principal Investigator — Riphah International University
Locations (1):
- Jinnah Hospital, gynae ward, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Paul J, Khanam S, Jain P. Comparative effect of Aerobic Training versus Plyometric Training among Young Obese Women with Poly Cystic Ovarian Syndrome. www ijmaes org.
- [Background] Yilmaz B, Vellanki P, Ata B, Yildiz BO. Metabolic syndrome, hypertension, and hyperlipidemia in mothers, fathers, sisters, and brothers of women with polycystic ovary syndrome: a systematic review and meta-analysis. Fertil Steril. 2018 Feb;109(2):356-364.e32. doi: 10.1016/j.fertnstert.2017.10.018. Epub 2018 Jan 11. PMID 29331234
- [Background] Flor-Rufino C, Barrachina-Igual J, Perez-Ros P, Pablos-Monzo A, Martinez-Arnau FM. Resistance training of peripheral muscles benefits respiratory parameters in older women with sarcopenia: Randomized controlled trial. Arch Gerontol Geriatr. 2023 Jan;104:104799. doi: 10.1016/j.archger.2022.104799. Epub 2022 Aug 29. PMID 36070636
- [Background] Crosignani PG, Colombo M, Vegetti W, Somigliana E, Gessati A, Ragni G. Overweight and obese anovulatory patients with polycystic ovaries: parallel improvements in anthropometric indices, ovarian physiology and fertility rate induced by diet. Hum Reprod. 2003 Sep;18(9):1928-32. doi: 10.1093/humrep/deg367. PMID 12923151
- [Background] Welt CK, Carmina E. Clinical review: Lifecycle of polycystic ovary syndrome (PCOS): from in utero to menopause. J Clin Endocrinol Metab. 2013 Dec;98(12):4629-38. doi: 10.1210/jc.2013-2375. Epub 2013 Sep 24. PMID 24064685
- [Background] Abraham Gnanadass S, Divakar Prabhu Y, Valsala Gopalakrishnan A. Association of metabolic and inflammatory markers with polycystic ovarian syndrome (PCOS): an update. Arch Gynecol Obstet. 2021 Mar;303(3):631-643. doi: 10.1007/s00404-020-05951-2. Epub 2021 Jan 13. PMID 33439300
- [Background] Repaci A, Gambineri A, Pasquali R. The role of low-grade inflammation in the polycystic ovary syndrome. Mol Cell Endocrinol. 2011 Mar 15;335(1):30-41. doi: 10.1016/j.mce.2010.08.002. Epub 2010 Aug 11. PMID 20708064
- [Background] Miranda-Furtado CL, Ramos FK, Kogure GS, Santana-Lemos BA, Ferriani RA, Calado RT, Dos Reis RM. A Nonrandomized Trial of Progressive Resistance Training Intervention in Women With Polycystic Ovary Syndrome and Its Implications in Telomere Content. Reprod Sci. 2016 May;23(5):644-54. doi: 10.1177/1933719115611753. Epub 2015 Nov 18. PMID 26586671